CLINICAL TRIAL: NCT01840722
Title: Brief Intervention for Rural Women at High Risk for HIV/HCV
Acronym: WISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Staton (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Michele Staton, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R01DA033866-02 (NIH); 5R01DA033866-02 (NIH)
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-08

CONDITIONS: Acquired Immune Deficiency Syndrome Virus; Hepatitis C; Drug Abuse
Keywords: HIV; HCV; Substance abuse; women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIDA Standard HIV Education (No Intervention): NIDA Standard HIV Education Participants in this condition will be given HIV education using NIDA standard pre and post-test counseling, HIV and HCV rapid testing, and an information packet on existing community drug abuse and HIV/HCV resources
- MI-based HIV Risk Reduction (Experimental): MI-based HIV Risk Reduction -- In addition to what is received in the HIV-Ed group, participants in this condition will also receive a CDC evidence-based brief intervention for high-risk women focused on an individualized plan for enhancing motivation to reduce risk behaviors and to use health and behavioral health services in the community.
  Interventions: Other: MI-based HIV Risk Reduction

INTERVENTIONS:
Other: MI-based HIV Risk Reduction — As the only MI-based intervention identified by the CDC as a best-practice model, the MI-HIV intervention has been shown to demonstrate positive outcomes for criminal justice-involved women randomly assigned to the intervention group for risky sexual activity and drug use with sustained behaviors through 9 months.
  Other Names: Motivational Interviewing for HIV Risk Reduction; Portland Women's Health Program
  Arms: MI-based HIV Risk Reduction

SUMMARY:
The overall aim of this study is to reduce risk behaviors and increase health and behavioral health service utilization among disadvantaged, drug-using rural women at high risk for HIV and HCV. This project has potential to make a significant contribution to science by providing knowledge about the health, risk behaviors, and service utilization of a vulnerable and understudied group of women during a time of emerging and significant public health risk in a rural Appalachian setting. Successful completion of the aims of this project will advance the delivery of a low-cost, potentially high impact intervention with implications for a number of other real world settings (such as criminal justice venues) where other disadvantaged high-risk drug users can be identified and targeted for intervention.

DETAILED DESCRIPTION:
Specific Aim 1: Compare the effectiveness of an evidence-based HIV risk reduction intervention (MI-HIV) to HIV Education (NIDA Standard) in reducing sex risk behaviors, injection practices, and drug use among a culturally unique sample of disadvantaged, drug-using rural women at high-risk for HIV and HCV. This aim will be accomplished through the random selection of high-risk rural women drug users from rural jails, screening and assessment for high-risk behavior, and random assignment to the HIV-Ed or MI-HIV intervention conditions. Follow-up interviews at 3, 6, and 12 months in the community post-release will examine changes in high-risk behavior. It is expected that MI-HIV participants will report significantly greater reductions in risky injection drug use practices, other drug use, and sex risk behaviors than women who participate in the HIV-Ed condition.

Specific Aim 2: Examine MI-HIV Intervention engagement as a predictor of community health and behavioral health service utilization (including drug treatment and mental health) at follow-up among disadvantaged, drug-using rural women at high risk for HIV and HCV. This aim will focus on community service utilization during the follow-up period by the intervention and education comparison group, and how health and behavioral health service utilization relates to patterns of HIV/HCV risk behavior. It is expected that MI-HIV participants will utilize more services due to increased motivation for treatment and treatment planning following the brief intervention.

ELIGIBILITY:
Inclusion Criteria:

* ASSIST score of 4+
* engagement in at least one sex risk behavior in the past 3 months
* willingness to participate in brief intervention sessions
* no evidence of cognitive impairment
* no evidence of active psychosis (currently experiencing hallucinations)
* no self-reported current symptoms of physical withdrawal from a recent episode of drug use
* incarceration period of 1 week - 3 months in order to complete intervention sessions

Exclusion Criteria:

* ASSIST score of <4
* no engagement in at least one sex risk behavior in the past 3 months
* not willing to participate in brief intervention sessions
* evidence of cognitive impairment
* evidence of active psychosis (currently experiencing hallucinations)
* self-reported current symptoms of physical withdrawal from a recent episode of drug use
* incarceration period of less than 1 week or greater than 3 months in order to complete intervention sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tindall, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Rural Appalachian Research Center, Hazard, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
N/A, individual participant data will not be made available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult women were randomly selected from three rural jails in Appalachia, screened, and interviewed face-to-face in a private room in the jail. Study eligibility included: 1) moderate risk of substance abuse based on the NIDA-ASSIST score of 4+ for any drug; 2) residing in Appalachia before incarceration; and 3) willingness to participate.
Pre-assignment Details: Of the 688 screened, 248 (36%) did not meet eligibility criteria due to: not being released during time frame (n=203), not engaging in risky sexual practices (n=15), not being from Appalachian (n=21), and not meeting NM-ASSIST criteria (n=9). 440 (64%) met criteria, but 40 were released prior to completing the baseline. The final N=400.
Period: Overall Study
Arm/Group | NIDA Standard HIV Education | MI-based HIV Risk Reduction
Started | 201 | 199
Completed | 201 | 130
Not Completed | 0 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIDA Standard HIV Education | MI-based HIV Risk Reduction | Total
Number analyzed (Participants) | 201 | 199 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 201 | 199 | 400
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (8.4) | 33.1 (8.1) | 32.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 199 | 400
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 200 | 197 | 397
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 201 | 199 | 400
Risky Sexual Behavior [Count of Participants; unit: Participants] — Ever Had Sex with a Partner in Exchange for Money, Drugs, Food, Shelter, Transportation, etc
  Participants | 84 | 90 | 174

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having Unprotected Casual Sex
Description: Had unprotected sex with a casual partner or when trading sex for money, drugs, etc in the past 6 months
Time Frame: 6 months
Population: Participants were lost to study attrition
Measure: Count of Participants; unit: Participants
Arm/Group | NIDA Standard HIV Education | MI-based HIV Risk Reduction
Number analyzed (Participants) | 181 | 184
Participants | 27 | 25

2. Secondary Outcome: Number of Participants Exchanging Sex
Description: Sex with a Partner in Exchange for Money, Drugs, Food, Shelter, Transportation, etc. in the past 6 months
Time Frame: 6 months
Population: Participants were lost to attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | NIDA Standard HIV Education | MI-based HIV Risk Reduction
Number analyzed (Participants) | 181 | 184
Participants | 9 | 8

3. Secondary Outcome: Number of Participants Recently Receiving Physical or Behavioral Health Treatment
Description: Is currently being treated for a physical or mental health problem OR has been in a substance use treatment program in the last 6 months
Time Frame: 6 months
Population: Participants were lost to study attrition.
Measure: Count of Participants; unit: Participants
Arm/Group | NIDA Standard HIV Education | MI-based HIV Risk Reduction
Number analyzed (Participants) | 181 | 184
Participants | 83 | 84

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for one year post-study enrollment.
Description: The definitions of adverse events in this study do not differ from clinicaltrials.gov definitions.
Arm/Group | NIDA Standard HIV Education | MI-based HIV Risk Reduction
All-Cause Mortality (participants affected / at risk) | 2/201 | 1/199
Serious Adverse Events (participants affected / at risk) | 2/201 | 1/199
Other Adverse Events (participants affected / at risk) | 0/201 | 0/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIDA Standard HIV Education (N=201) | MI-based HIV Risk Reduction (N=199)
Participant death (Investigations) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-03-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT01840722/Prot_000.pdf